CLINICAL TRIAL: NCT06849583
Title: Comparison of the Effects of Preoperative Anesthesia Evaluation on Preoperative Anxiety Using Anxiety Scales and Evaluation of Patient Satisfaction; Prospective Study
Brief Title: Comparison of the Effects of Preoperative Anesthesia Evaluation on Preoperative Anxiety Using Anxiety Scales and Evaluation of Patient Satisfaction
Status: Enrolling by invitation | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2019.02.31
Record Dates: First submitted 2025-02-14; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Evaluation; Preoperative Anxiety; STAI; Visual Analogy Scala; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm Preinterview
- Arm Postinterview

SUMMARY:
To measure the degree of preoperative anxiety with the STAIT, APAIS and VAS anxiety scales before and after the preoperative anesthesia evaluation in patients who applied for preoperative anesthesia evaluation for elective surgical procedures and to investigate prospectively the effect of the preoperative anesthesia interview on anxiety and to evaluate patient satisfaction.

DETAILED DESCRIPTION:
Anxiety is one of the diseases that has recently attracted worldwide attention and seriously affects daily life. Preoperative anxiety is a significant problem for patients because it causes physical problems as well as emotional and psychiatric disorders. It negatively affects surgery, anesthesia and postoperative recovery and is seen in 60-80% of patients scheduled for surgery. Most patients experience varying degrees of anxiety and fear before surgery. This anxiety and fear may depend on the type of anesthesia, as well as the patient's previous experiences, personality traits, concerns about the surgical procedure and postoperative pain. Preoperative anxiety causes difficulties in anesthesia induction, autonomic fluctuations and increased anesthetic requirements, and has been associated with increased pain, nausea and vomiting, prolonged recovery and prolonged hospitalization in the postoperative period. Anxious patients encounter complications in the perioperative period at a higher incidence. Anxiety assessment is important because anxious patients' responses to anesthesia and analgesia are different than those of non-anxious patients. For this purpose, anxiety can be assessed in many ways, directly by measuring plasma cortisol and urinary catecholamines, and indirectly by measuring pulse and blood pressure.

Preoperative anxiety begins when the surgical procedure is planned and reaches its maximum intensity at hospital admission. Correct management of fear and anxiety is achieved by a better preoperative assessment and information provided by anesthesiologists. Therefore, anxious patients should be routinely identified during preoperative assessment.

In practice, there are different anxiety scales that can be used to define patient anxiety within a limited time. Many documents have been reported on the assessment of preoperative anxiety. One of these is the State-Trait Anxiety Inventory (STAI) scale, which is the most widely used test for assessing anxiety at a specific time. In addition, the Amsterdam Preoperative Anxiety and Information Scale (APAIS), which is simpler and less time-consuming to apply, was developed to measure anxiety and desire for information related to anesthesia and surgery, and its usability and correlation with STAI were investigated. The Visual Analog Scale (VAS) (range 0-100 mm) is an alternative scale used to assess anxiety, consisting of a 100 mm line; zero on the left indicates no anxiety, while 100 mm on the right indicates extreme anxiety.

Previous studies have identified that patients feel anxious before elective surgery, but studies investigating the effect of preassessment clinics (PACs) on anxiety levels have been limited to the use of patient information literature or multimedia rather than the preoperative anesthesia consultation process. Since PACs have the potential to provide patients with a better understanding of their anesthesia and surgery, they have the potential to reduce anxiety.

The aim of this study was to measure the degree of preoperative anxiety in patients presenting to our anesthesia outpatient clinic before and after the preoperative anesthesia assessment using the STAIT, APAIS and VAS anxiety scales, and to investigate the effect of the preoperative anesthesia interview on anxiety and to evaluate patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo elective surgery
* Sufficient language skills for the interview
* Ages 16-85
* ASA I - III
* Patients who apply to the anesthesia clinic for anesthesia evaluation

Exclusion Criteria:

* Patients under the age of 16
* Patients who do not consent
* Those who do not have sufficient language skills
* Those with mental and/or psychiatric disorders
* Emergency and/or ASA-IV patients
* Those with a history of sedative drug use

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was prepared as an observational prospective study. Patients between the ages of 16-85 who apply for preoperative anesthesia evaluation for elective surgical procedures by an anesthesiologist in the Anesthesia Polyclinic will be invited to the study. The effect of preoperative anesthesia evaluation on preoperative anxiety will be investigated with the help of anxiety scales.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety scales (State- Trait Anxiety Inventory , Amsterdam Preoperative Anxiety and Information Scale , Visuel Analog Skala ) | Three days from registration to completion and evaluation of all patient questionnaires
  To measure the degree of preoperative anxiety in adult patients admitted to our anesthesia clinic using the STAIT, APAIS and VAS anxiety scales before and after preoperative anesthesia evaluation and to prospectively investigate the effect of the preoperative anesthesia interview on anxiety and to evaluate patient satisfaction.The Visual Analog Scale (VAS) (range 0-100 mm) is an alternative scale used in the assessment of anxiety, consisting of a 100 mm line; zero on the left indicates no anxiety, while 100 mm on the right indicates extreme anxiety. In the Spielberger State-Trait Anxiety Inventory (STAI), patients with a score of 45 and above will be considered highly anxious (mild ≤39, moderate = 40-45, severe ≥46). In the Amsterdam Preoperative Anxiety and Information Scale (APAIS), patients with an APAIS-A score greater than 10 will be considered highly anxious. Patients with an APAIS-B score of 5 and above will be considered to have a need for information.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)